CLINICAL TRIAL: NCT06149468
Title: CAP48 Medical Research Project: Autism Spectrum Disorders in Children and Adolescents
Brief Title: CAP48 - Autism in Children and Adolescents
Acronym: CAP48-ASD
Status: Recruiting | Type: Observational
Sponsor: Université Catholique de Louvain (Other)
Collaborators: Université Libre de Bruxelles (Other); Université de Namur (Unknown); University of Mons (Other); Université de Liège (Other)
Responsible Party: Sponsor
Other Study IDs: CAP48 - TSA
Record Dates: First submitted 2023-11-20; First posted 2023-11-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ASD group: child/adolescent (under 18 years of age) applying to an autism reference center or being followed up in an autism reference center
  Interventions: Other: inclusion in the register

INTERVENTIONS:
Other: inclusion in the register — socio-demographic data collection and proposed therapy

SUMMARY:
Evaluation and follow-up of children diagnosed with an autism spectrum disorder in French-speaking Belgium in order to optimize diagnostic protocols, the quality of care required and its accessibility, and to determine the impact of an autism spectrum disorder on schooling, family and society.

DETAILED DESCRIPTION:
The aims of the research project:

* To collect a wide range of data in order to improve knowledge of children with autism spectrum disorder (ASD) in French-speaking Belgium by prospectively including all children and adolescents making a request to the centres of reference. The creation of a common database will make it possible to collect general socio-demographic, geographical and epidemiological data, to characterise the different profiles and to accurately monitor developmental trajectories.
* Evaluate the feasibility and practical implementation of the treatment proposed following a diagnosis of ASD in a child.
* Implement protocols to improve the quality of care for beneficiaries.
* To enable the development of fundamental research protocols. Many questions remain unanswered about the genetic, neuro-cognitive and linguistic characteristics of autism. Only rigorous studies carried out on large, carefully defined samples can advance research.
* Increase public knowledge and understanding of the ASD.

ELIGIBILITY:
Inclusion Criteria:

* children/adolescents (under 18 years of age) who apply to an autism reference center or who are followed up in an autism reference center from French-speaking region of Belgium.

Exclusion Criteria:

* refusal by the family to allow their child's data to be included in the database.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children/adolescents (under 18 years of age) who apply to an autism reference center or who are followed up in an autism reference center.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Creation of an ADS register | Throughout the entire study, approximately during 5 years
  creation of a common ASD register to collect general sociodemographic, geographic and epidemiological data, characterize the different patient profiles and accurately track development trajectories

SECONDARY OUTCOMES:
Feasability assessment | Throughout the entire study, approximately during 5 years
  Evaluate the feasibility and practical realization of the proposed care following a diagnosis of ASD in a child and implement protocols to improve the quality of therapy.
Protocols development | Throughout the entire study, approximately during 5 years
  Enable the development of fundamental research protocols: genetic, neurocognitive and linguistic
Schooling evaluation | Throughout the entire study, approximately during 5 years
  Evaluate the schooling of children with ASD of all ages

CONTACTS AND LOCATIONS:
Overall Officials: Marine Houssa, PhD, Study Chair — Université Catholique de Louvain
Locations (1):
- UCLouvain, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No